CLINICAL TRIAL: NCT06997133
Title: Sucralose as a Way to Enhance Regulatory T Cells: The Sweet Trial
Brief Title: Sucralose as a Way to Enhance Regulatory T Cells
Acronym: SWEET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caroline Lamarche (Other)
Collaborators: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor-Investigator, Caroline Lamarche, Principal Investigator, clinical assistant professor, Ciusss de L'Est de l'Île de Montréal
Organization: Ciusss de L'Est de l'Île de Montréal (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2025-3912
Record Dates: First submitted 2024-12-20; First posted 2025-05-30 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteer
Keywords: sucralose; immune system; regulatory T cells; metabolomic
MeSH Terms: interventions — trichlorosucrose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Starting with placebo - washout - sucralose. (Placebo Comparator): This group will start with a placebo (4 weeks) , then will have a washout period (2 weeks) and then will test sucralose (4 weeks)
  Interventions: Dietary Supplement: sucralose; Other: Placebo
- Starting with sucralose - washout - placebo. (Active Comparator): This group will start with sucralose (4 weeks) , then will have a washout period (2 weeks) and then will test the placebo (4 weeks)
  Interventions: Dietary Supplement: sucralose; Other: Placebo

INTERVENTIONS:
Dietary Supplement: sucralose — Encapsulated sucralose po BID
Other: Placebo — Encapsulated lactose po bid

SUMMARY:
Title: Taking the SWEET approach to protect the transplanted kidney.

Background: Kidneys are essential organs in our body. When they do not work, patients require machines to help them or receive a new kidney from a donor (transplantation) to survive. Thus far, transplantation is the best treatment. However, the immune system will recognize the new kidney as foreign and try to destroy it, which is called kidney rejection. To prevent rejection, patients with kidney transplants depend on drugs to suppress the immune system. However, these drugs have many side effects, including the risk of infection, cancer, and diabetes.

The immune system is made of many different types of cells. One cell type in particular is T cells that, when kept unchecked, will attack the kidney transplant. However, there is a small subset of these T cells called regulatory T cells (Tregs) that police the immune system and aid in accepting the new kidney. Current ways to increase these police cells (Tregs) after a transplant are expensive and not widely available. Therefore, there is a need to find a better and more accessible way to increase Treg numbers after a transplant to increase the longevity of the newly transplanted kidney.

What we eat is critical in shaping the immune system. Artificial sweeteners, like sucralose (found in Splenda), are often used as a sugar substitute. They are low in calories and safe to consume. However, recent studies suggest they may have unexpected effects on the body. Research in mice has shown that sucralose impacts the immune system. Specifically, the investigators have found that it could suppress T cells that could cause kidney rejection while increasing the Tregs (the police).

Given these findings, the investigators hypothesize that sucralose could be beneficial in conditions where dampening the immune system is desirable, such as in the case of transplantation. By boosting Tregs and reducing the anti-transplant T cells, sucralose may help to protect against organ rejection.

Purpose: The goal of this study is thus to test whether sucralose can safely and effectively modulate the immune system in humans.

Method: The investigator propose to test the impact of sucralose on the immune system. This pilot study will test the effect of sucralose in 10 healthy volunteers. The participants will take sucralose or placebo as a pill twice daily for a month. Healthy volunteers will then stop for a two weeks (washout period). After the washout period, the volunteers on sucralose will switch to placebo, while the placebo group will switch to sucralose pills for one more months. The investigators will take blood samples at the beginning, after one month, after the washout and at the end of the study to study how the immune system changes.

Anticipated outcomes: The investigators expect that sucralose will impact the immune system and increase the number of regulatory T cells.

Relevance to patient/community: Artificial sweeteners are commonly used in the food and pharmaceutical industries. However, their impact on the immune system has not been thoroughly investigated in humans.

Conclusion: Kidney transplantation is the most effective treatment for kidney failure, but the immune system's rejection of the transplanted organ remains a major challenge. Current immunosuppressive drugs used to prevent rejection have significant side effects, underscoring the need for safer alternatives. The investigator research suggests that sucralose, a widely used artificial sweetener, may offer a novel solution by increasing the good T cells (Tregs) and reducing harmful T cells that contribute to rejection. This pilot study will explore sucralose's potential to modulate the immune system in humans, potentially leading to improved transplant outcomes and broader implications for immune regulation.

ELIGIBILITY:
Inclusion Criteria:

* Body weight comparable to average reported in Canada

Exclusion Criteria:

* Past medical history of autoimmune disease
* The use of any regular medication except contraceptive pills
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Regulatory T cells | After 4 weeks on sucralose and placebo.
  Change in % regulatory T cells on total CD4+ T cells compared to baseline

SECONDARY OUTCOMES:
T cell cytokine production (TNFa, IFNy, IL2) | 4 weeks compared to baseline on either placebo or sucralose
  % cytokine production o CD4+ and CD8+ T cells
Frequency of immune populations in the blood (CD4+, CD8+, NK, B cells, CD11b myeloid cells) | 4 weeks compared to baseline on either sucralose or placebo
  % of CD45+ cells (total immune marker)
Frequency of CD4+ T cells lineages | 4 weeks compared to baseline on sucralose or placebo
  % RORyt, T-bet, GATA3 on CD4+ T cells
Frequency of naive, central and effector memory or terminally differentiated CD4+ and CD8+ T cells | 4 weeks compared to baseline on both sucralose or placebo
  % of CD62L+CD45RA+CD45RO- (naive), CD62L+CD45RO+CD44+CD45RA- (central memory), CD62L-CD45RA-CD45RO+CD44+ (effector memory) and CD62L-CD45RA+CD45RO (terminally differentiated cells) on both CD4+ and CD8+ T cells

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche de l'Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No